CLINICAL TRIAL: NCT04512755
Title: AIMS Medical Outcomes Study
Acronym: AMOS
Status: Recruiting | Type: Observational
Sponsor: Advanced Integrative Medical Science Institute (Other)
Responsible Party: Sponsor
Other Study IDs: AMOS
Record Dates: First submitted 2020-07-30; First posted 2020-08-14 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Mental Health Issue; PTSD; Pain; Chronic Pain; Chronic Disease
Keywords: Naturopathic Oncology; Integrative Medicine; Integrative Psychiatry; Integrative Physical Medicine and Rehabilitation; Integrative Palliative Care Medicine; Serious Illness; Life Threatening Illness
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Pain; Chronic Pain; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This epidemiologic research is being conducted as an observational prospective case series outcomes study of the use of advanced integrative specialty medical care and its effect on adult and pediatric patients with chronic or serious illnesses or mental health disorders.

DETAILED DESCRIPTION:
There is growing interest in providing integrative medical care in conjunction with specialty medical care to expand the reach of integrative care to more chronically and seriously ill patient populations. At the AIMS Institute, the core specialties are naturopathy, palliative care, psychiatry, physiatry, and naturopathic oncology practiced via coordinated, team-based care by allopathic medical and psychiatric specialists, psychotherapists, specialized naturopathic physicians, advanced practice nurses, and targeted health educators, with the majority of care covered by insurance. Additionally incorporated are novel 'advanced' approaches, such as drug-assisted psychotherapy, medical cannabis education, sympathetic blocks, and some intravenous therapies.

This is an uncontrolled, prospective case series outcomes study of health-related quality of life outcomes in patients who receive care at AIMS Institute. A clinic-wide chart audit of patient characteristics and outcomes will be conducted prior to the start of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in the study will meet the following criteria:

  1. A new patient coming in for a first office call (FOC) or first consultation via telemedicine with an AIMS physician or advanced practice provider;
  2. An established patient;
  3. If over 18 years of age are able to understand study design adequately and provide signed informed consent to enrollment;
  4. If younger than 18 years of age informed consent from a parent or guardian who is able to understand the study design adequately and provide signed informed consent for the pediatric patient.

Exclusion Criteria:

* Ineligible participants:

  1. Cannot read or understand English well enough to read and sign the consent form and complete the questionnaires;
  2. Unwilling to participate in the AIMS Institute observational study.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients who seek care at AIMS Institute and meet inclusion/exclusion criteria are eligible to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Health Related Quality of Life | 5 Years
  Measure quality of life using GAD-7, PHQ-9, and short form questionnaire.

SECONDARY OUTCOMES:
Treatment | 5 Years
  Describe treatments prescribed and provided by AIMS Institute physicians abstracted from chart review.

CONTACTS AND LOCATIONS:
Overall Officials: Therry Eparwa, DNP, FNP-BC, Principal Investigator — AIMS Institute; Sunil K Aggarwal, MD, PhD, Study Director — AIMS Institute; Leanna J Standish, ND, PhD, LAc, Study Director — AIMS Institute
Locations (1):
- AIMS Institute, Seattle, Washington, United States

REFERENCES:
- [Background] De Lima L, Bennett MI, Murray SA, Hudson P, Doyle D, Bruera E, Granda-Cameron C, Strasser F, Downing J, Wenk R. International Association for Hospice and Palliative Care (IAHPC) List of Essential Practices in Palliative Care. J Pain Palliat Care Pharmacother. 2012 Jun;26(2):118-22. doi: 10.3109/15360288.2012.680010. PMID 22764847
- [Background] Stjernsward, J. & Clark, D. (2005). Palliative medicine: a global perspective. In Doyle, D., Hanks, G., Cherny, N., & Calman, K. (Eds.). Oxford textbook of palliative medicine (3rd ed., pp. 1197-224). Oxford University Press.
- [Background] Bercovitz A, Sengupta M, Jones A, Harris-Kojetin LD. Complementary and alternative therapies in hospice: The national home and hospice care survey: United States, 2007. Natl Health Stat Report. 2011 Jan 19;(33):1-20. PMID 25585442
- [Background] Leskowitz E. (2002) Complementary and alternative medicine in rehabilitation. Churchill Livingstone.
- [Background] Monti, D.A. & Newberg, A.B. (2018). Integrative psychiatry and brain health (2nd ed.) Weil Integrative Medicine Library, Oxford University Press.
- [Background] Scotton, B.W., Chinen, A.B., &Battista, J.R. (Eds.). (1996). Textbook of transpersonal psychiatry and psychology. Basic Books.
- [Background] Association of Accredited Naturopathic Medical Colleges. (2019). Naturopathic medicine: Become the doctor you want to have. [Whitepaper]. Association of Accredited Naturopathic Medical Colleges. Retrieved May 13, 2020 from: https://aanmc.org/wp-content/uploads/2019/02/Naturopathic-Medicine-White-Paper.pdf
- [Background] Standish, L.J. & Aggarwal, S.K. (2019). Advanced integrative oncology treatment for adult and pediatric patients with cancer: A prospective outcomes study. AIMS Institute Clinical Study Protocol.
- [Background] Wolfson, P. & Hartelius, G. (Eds). (2016). The ketamine papers: Science, therapy, and transformation. Multidisciplinary Association for Psychedelic Studies.
- [Background] Ghebreyesus, Tedros Adhanom. (2019, January 24). Tedros Adhanom Ghebreyesus to António Guterres. World Health Organization. Retrieved from https://www.who.int/medicines/access/controlled-substances/UNSG_letter_ECDD41_recommendations_cannabis_24Jan19.pdf
- [Background] Cyr C, Arboleda MF, Aggarwal SK, Balneaves LG, Daeninck P, Neron A, Prosk E, Vigano A. Cannabis in palliative care: current challenges and practical recommendations. Ann Palliat Med. 2018 Oct;7(4):463-477. doi: 10.21037/apm.2018.06.04. Epub 2018 Jun 28. PMID 30180728
- [Background] Wolever RQ, Abrams DI, Kligler B, Dusek JA, Roberts R, Frye J, Edman JS, Amoils S, Pradhan E, Spar M, Gaudet T, Guarneri E, Homel P, Amoils S, Lee RA, Berman B, Monti DA, Dolor R. Patients seek integrative medicine for preventive approach to optimize health. Explore (NY). 2012 Nov-Dec;8(6):348-52. doi: 10.1016/j.explore.2012.08.005. PMID 23141791
- [Background] Abrams DI, Dolor R, Roberts R, Pechura C, Dusek J, Amoils S, Amoils S, Barrows K, Edman JS, Frye J, Guarneri E, Kligler B, Monti D, Spar M, Wolever RQ. The BraveNet prospective observational study on integrative medicine treatment approaches for pain. BMC Complement Altern Med. 2013 Jun 24;13:146. doi: 10.1186/1472-6882-13-146. PMID 23800144
- [Background] Edman JS, Roberts RS, Dusek JA, Dolor R, Wolever RQ, Abrams DI. Characteristics of cancer patients presenting to an integrative medicine practice-based research network. Integr Cancer Ther. 2014 Sep;13(5):405-10. doi: 10.1177/1534735414537876. Epub 2014 Jun 9. PMID 24913179
- [Background] Dusek JA, Abrams DI, Roberts R, Griffin KH, Trebesch D, Dolor RJ, Wolever RQ, McKee MD, Kligler B. Patients Receiving Integrative Medicine Effectiveness Registry (PRIMIER) of the BraveNet practice-based research network: study protocol. BMC Complement Altern Med. 2016 Feb 4;16:53. doi: 10.1186/s12906-016-1025-0. PMID 26846166
- [Background] Ameli R, Sinaii N, Luna MJ, Cheringal J, Gril B, Berger A. The National Institutes of Health measure of Healing Experience of All Life Stressors (NIH-HEALS): Factor analysis and validation. PLoS One. 2018 Dec 12;13(12):e0207820. doi: 10.1371/journal.pone.0207820. eCollection 2018. PMID 30540764